CLINICAL TRIAL: NCT04987294
Title: A Randomized, Double-Blind, Placebo-Controlled Study of ALLN-346 (Engineered Urate Oxidase) in Hyperuricemic Subjects With Gout and Mild to Moderate Chronic Kidney Disease
Brief Title: Phase IIa Study of ALLN-346 (Engineered Urate Oxidase) in Subjects With Hyperuricemia, Gout and Chronic Kidney Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company Financing
Sponsor: Allena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALLN-346-202
Record Dates: First submitted 2021-07-26; First posted 2021-08-03 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Hyperuricemia; Gout; Chronic Kidney Diseases
MeSH Terms: conditions — Hyperuricemia; Gout; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 2:1 to receive ALLN-346 or placebo.
Who Masked: Participant, Investigator
Masking Description: Subjects, Investigators and laboratories involved in the conduct of the study will be blinded to subject treatment assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALLN-346 (Engineered Urate Oxidase) (Experimental): ALLN-346 is novel urate oxidase provided as capsules for oral administration. ALLN-346 will be administered as 5 capsules thrice daily (15 capsules per day total) to each of two subject cohorts based on estimated glomerular filtration rate (eGFR). Treatment Period is 14 Days.
  Interventions: Drug: ALLN-346
- Placebo (Placebo Comparator): Matching placebo capsules for oral administration. Placebo capsules will be administered as 5 capsules thrice daily (15 capsules per day total) to each of two subject cohorts based on estimated glomerular filtration rate (eGFR). Treatment Period is 14 Days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALLN-346 — ALLN-346 (Engineered Urate Oxidase) is an orally administered, novel urate oxidase; provided as capsules for oral administration
  Other Names: Engineered urate oxidase
  Arms: ALLN-346 (Engineered Urate Oxidase)
Drug: Placebo — Matched placebo capsules are similar in weight and appearance to the ALLN-346 capsules
  Other Names: Matching placebo capsule
  Arms: Placebo

SUMMARY:
The purpose of this Phase IIa study is to evaluate the safety, tolerability and pharmacodynamics of ALLN-346 in subjects with hyperuricemia and gout, and with mild to moderate chronic kidney disease.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled parallel group, multi-center phase II clinical study or orally administered ALLN-346 in subjects with hyperuricemia, gout and mild to moderate chronic kidney disease over a two-week period. Subjects will be enrolled in two cohorts based on estimated glomerular filtration rate (eGFR).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 to 70 years
* Serum UA level ≥ 8.0 mg/dL at Screening (hyperuricemia)
* Meets 2015 American College of Rheumatology (ACR)/EULAR criteria for gout
* Screening eGFR of ≥60 - <90 mL/minute/1.73 m2 for Cohort A and ≥30 - <60 mL/minute/1.73 m2 for Cohort B.
* Concomitant medications stable for a minimum of 4 weeks prior to and during Screening
* Body Mass Index (BMI) ≥ 18 and ≤ 40 kg/m2, inclusive, at screening
* Not pregnant, not capable of pregnancy, not nursing, and agrees to use an effective method of contraception; males subjects must agree to abstain from sperm donation

Exclusion Criteria:

* Currently taking any oral urate-lowering medication within 2 weeks prior to Screening
* Prior uricase therapy or exposure to recombinant uricase, such as Rasburicase or Pegloticase
* Gout flare requiring treatment within 14 days prior to or during Screening
* Clinically significant finding during Screening, any ongoing clinically significant illness requiring a clinically significant intervention or change in management within 4 weeks prior to or during Screening
* History of GI surgery, including gastric sleeve, Roux-en-Y or gastric banding (unless gastric band removed for a minimum of 12 months prior to Screening
* Received treatment with or exposure to an Investigational drug or device within 30 days - prior to or during Screening
* Prior dosing in ALLN-346 clinical study
* Per Investigator judgment, is not an ideal clinical study candidate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | 42 days
  Treatment emergent adverse events

SECONDARY OUTCOMES:
Serum Urate | 14 Days
  Serum urate [mg/dL]

CONTACTS AND LOCATIONS:
Overall Officials: C Tosone, MS, RAC, Study Director — Allena Pharmaceuticals
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Syed Research Consultants, LLC, Muscle Shoals, Alabama
  - Syed Research Consultants, LLC, Sheffield, Alabama
  - Orthopedic Physicians Alaska, Anchorage, Alaska
  - Allameh Medical Corporation, Mission Viejo, California
  - Eastern Research, Inc., Hialeah, Florida
  - Best Quality Research, Inc., Hialeah, Florida
  - New Generation of Medical Research, Hialeah, Florida
  - Kendall South Medical Center, Inc., Miami, Florida
  - The Center of Rheumatology and Bone Research, Wheaton, Maryland
  - Elite Clinical Research, LLC, Jackson, Mississippi
  - NY Total Medical Care, PC, Brooklyn, New York
  - Burke Primary Care, Morganton, North Carolina
  - Summit research Group, LLC, Stow, Ohio
  - Northeast Clinical Research Center, LLC, Bethlehem, Pennsylvania
  - P&I Clinical Research, LLC, Lufkin, Texas
  - Briggs Clinical Research, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No